CLINICAL TRIAL: NCT02540473
Title: Fostering Resilience: An Intervention for Women Physicians at Risk for Burnout
Brief Title: Fostering Resilience in Physician Moms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Cynthia M. Stonnington, M.D., Associate Professor of Psychiatry, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-009196
Record Dates: First submitted 2015-08-28; First posted 2015-09-04 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Stress, Psychological
Keywords: Resilience
MeSH Terms: conditions — Stress, Psychological | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group therapy (Experimental): 12 week manualized group therapy (one hour per week)
  Interventions: Behavioral: Manualized Therapy
- Control Group (Other): Participants get one hour of time away from patient care/duties to do as they wish.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Manualized Therapy — Relational psychotherapy mothers
  Arms: Group therapy
Behavioral: Control Group — one hour of free time to do with as they wish
  Arms: Control Group

SUMMARY:
Physicians in general are at risk for burnout, and this risk is heightened among women, particularly mothers. In a randomized design, central hypotheses in this study are that mothers who attend our 12-week Relational Psychotherapy Mothers Group (RPMG) intervention will show significantly greater decreases in stress, depression, burnout, and associated risk biomarker indices, as compared to comparison controls (who would meet in unstructured gatherings, for an hour a week for 12 weeks). Additionally the investigators hypothesize that the gains would be maintained three months after the intervention is completed.

ELIGIBILITY:
Inclusion of Women and Minorities:

* This study will be restricted to women physician mothers, who are the target of the manualized RPMG program.
* The study will not use race or ethnicity as a basis for selecting subjects.

Inclusion of Children:

* This study does not include children.

Exclusion criteria

* Participation in this study is open to all Mayo physician mothers with a child under the age of 18 years.
* As in past RPMG trials, the only exclusion criteria are if mothers were to indicate active suicidality, or meet criteria for psychoses, during initial assessments or during participation in this study.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
level of depression | Baseline to 3 months
  Beck Depression Inventory

SECONDARY OUTCOMES:
biomarker of stress | Baseline to 3 months
  C-reactive protein
biomarker of stress | Baseline to 3 months
  nerve-growth factor
Professional functioning | Baseline to 3 months
  The Maslach Burnout Inventory
perceived social support | Baseline to 3 months
  Quality of Social Support Scale
Parenting stress | Baseline to 3 months
  Parenting Stress Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Stonnington, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860
- [Derived] Luthar SS, Curlee A, Tye SJ, Engelman JC, Stonnington CM. Fostering Resilience among Mothers under Stress: "Authentic Connections Groups" for Medical Professionals. Womens Health Issues. 2017 May-Jun;27(3):382-390. doi: 10.1016/j.whi.2017.02.007. Epub 2017 Apr 14. PMID 28410972